CLINICAL TRIAL: NCT01315795
Title: An Open-label, Phase II Clinical Study to Evaluate the Efficacy and Safety of Lanreotide Autogel 90mg Every 4 Weeks in the Treatment of Symptomatic Polycystic Liver Disease, Including a Dose Escalation at Month 6 to Lanreotide Autogel 120mg for Non Responders
Brief Title: Lanreotide Autogel in the Treatment of Symptomatic Polycystic Liver Disease
Acronym: LOCKCYST
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Principal Investigator, Dr Frederik Temmerman, Professor Dr Frederik Nevens, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-024604-10
Record Dates: First submitted 2011-01-11; First posted 2011-03-15 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Polycystic Liver Disease
Keywords: polycystic liver disease
MeSH Terms: conditions — Polycystic liver disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Symptomatic polycystic liver disease (PCLD) patients (Experimental): Symptomatic polycystic liver disease (PCLD) patients
  Interventions: Drug: Lanreotide Autogel 90 mg and 120 mg

INTERVENTIONS:
Drug: Lanreotide Autogel 90 mg and 120 mg — administration of lanreotide sc every 4 weeks (28 days)

SUMMARY:
An open-label, Phase II clinical study to evaluate the efficacy and safety of lanreotide autogel 90mg every 4 weeks in the treatment of symptomatic polycystic liver disease, including a dose escalation at month 6 to lanreotide autogel 120mg for non responders.

ELIGIBILITY:
Inclusion Criteria:

* Liver volume ≥ 4 liter
* ≥ 20 liver cysts
* Symptomatic patients defined as at least 2 out of 5 of the following symptoms related to mass effect irrespective of the intensity:

  * Abdominal distention perceived as uncomfortable
  * Frequent abdominal pain
  * Early satiety
  * Nausea (with the inclusion of dyspeptic complaints)
  * Dyspnea
* Diagnosed with ADPKD or ADPLD
* Male and female patients of 18 years and older
* Written informed consent

Exclusion Criteria:

* Creatinine clearance < 20 ml/min
* Patient who underwent a kidney transplant and received variable doses of immunosuppressive therapy and/or present signs of rejection in the past year
* Hormonal replacement therapy
* Hormonal contraception
* Pregnant or lactating
* Presenting with an uncontrolled disease (other than ADPKD/ADPLD)
* Planned to undergo any surgery of the liver during study participation
* Planned to undergo any surgery of the KIDNEY during study participation (ADPKD patients only)
* Patients with known allergies to somatostatin or its analogues or any of its components
* Patients who received somatostatin analogues in the 6 months preceding study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Reduction of total liver volume after 6 months of treatment measured by means of CT-scan. | 6 months
  Reduction of total liver volume after 6 months measured by means of CT-scan.
Reduction of total liver volume after 12 months of treatment by means of CT-scan | 12 months
  Reduction of total liver volume after 12 months of treatment by means of CT-scan
Reduction of total liver volume after 18 months of treatment by means of CT-scan | 18 months
  Reduction of total liver volume after 18 months of treatment by means of CT-scan

SECONDARY OUTCOMES:
Measurement of total liver and kidney volumes and cyst volumes at baseline. | Baseline
  Reduction of total liver volume Reduction of liver cyst volume Additonal reduction of total liver volume in the non responder group. Additonal reduction of liver cyst volume in the non responder group.
  % of patients with liver reduction > 100 ml in the non responder group. Reduction of total kidney volume (ADPKD patients only) after 6 months, 1 year and 18 months
Measurement of total liver and kidney volumes and cyst volumes after 6 months of treatment by means of CT scan | 6 months
  Reduction of total liver volume Reduction of liver cyst volume Additonal reduction of total liver volume in the non responder group. Additonal reduction of liver cyst volume in the non responder group.
  % of patients with liver reduction > 100 ml in the non responder group. Reduction of total kidney volume (ADPKD patients only) after 6 months, 1 year and 18 months
Measurement of total liver and kidney volume and cyst volume after 12 months of treatment by means of CT scan. | 12 months
  Reduction of total liver volume Reduction of liver cyst volume Additonal reduction of total liver volume in the non responder group. Additonal reduction of liver cyst volume in the non responder group.
  % of patients with liver reduction > 100 ml in the non responder group. Reduction of total kidney volume (ADPKD patients only) after 6 months, 1 year and 18 months
Measurement of total liver and kidney volumes and cyst volumes after 18 months of treatment by means of CT scan | 18 months
  Reduction of total liver volume Reduction of liver cyst volume Additonal reduction of total liver volume in the non responder group. Additonal reduction of liver cyst volume in the non responder group.
  % of patients with liver reduction > 100 ml in the non responder group. Reduction of total kidney volume (ADPKD patients only) after 6 months, 1 year and 18 months
Assessment of quality of life at baseline | baseline
  Assessment of quality of life at baseline
Assessment of quality of life after 6 months of treatment | 6 months
  Assessment of quality of life after 6 months of treatment
Assessment of quality of life after 12 months of treatment | 12 months
  Assessment of quality of life after 12 months of treatment
Assessment of quality of life after 18 months of treatment | 18 months
  Assessment of quality of life after 18 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Nevens, MD, PhD, Principal Investigator — UZ Leuven, Gasthuisberg
Locations (1):
- UZ Leuven, Gasthuisberg, Leuven, Provincie Vlaams-Brabant, Belgium

REFERENCES:
- [Result] van Keimpema L, Nevens F, Vanslembrouck R, van Oijen MG, Hoffmann AL, Dekker HM, de Man RA, Drenth JP. Lanreotide reduces the volume of polycystic liver: a randomized, double-blind, placebo-controlled trial. Gastroenterology. 2009 Nov;137(5):1661-8.e1-2. doi: 10.1053/j.gastro.2009.07.052. Epub 2009 Jul 29. PMID 19646443
- [Derived] Temmerman F, Ho TA, Vanslembrouck R, Coudyzer W, Billen J, Dobbels F, van Pelt J, Bammens B, Pirson Y, Nevens F. Lanreotide Reduces Liver Volume, But Might Not Improve Muscle Wasting or Weight Loss, in Patients With Symptomatic Polycystic Liver Disease. Clin Gastroenterol Hepatol. 2015 Dec;13(13):2353-9.e1. doi: 10.1016/j.cgh.2015.05.039. Epub 2015 Jun 12. PMID 26073493
- See also: Lanreotide reduces the volume of polycystic liver: a randomized, double-blind, placebo-controlled trial. — http://www.ncbi.nlm.nih.gov/pubmed/19646443